CLINICAL TRIAL: NCT01572870
Title: Duplication in CHIT1 Gene and the Risk for Aspergillus Lung Disease in CF Patients
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 450-10 CTIL; Chit 1
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis; Chit1
Keywords: Chit1; Cystic Fibrosis; Allergic Bronchopulmonary Aspergillosis (ABPA); Aspergillus
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- No ABPA nor Aspergillus infection: CF patients who had neither ABPA nor Aspergillus infection in the past (the control group)
- persistent Aspergillus infection, without ABPA: CF patients with persistent Aspergillus infection, without ABPA.
- Current or past ABPA infection: CF patients with current or past ABPA

SUMMARY:
Title: Duplication in Chitotriosidase (CHIT1) Gene and the Risk for Aspergillus Lung Disease in CF Patients.

Aim: To evaluate the link between CHIT1 duplication in CF patients and the predisposition to ABPA or persistent Aspergillus infection.

Patients: 40 CF patients. Design: Observational, single visit. Methods: All patients will be assessed for pulmonary function tests (PFT), sputum cultures, and blood tests for: CHIT1 duplication, immunoglobulin E (IgE) and Eosinophils levels. Part of the patients will be assessed for RAST, skin prick test.

Primary outcome measure is the difference in CHIT1 genotyping between the groups.

DETAILED DESCRIPTION:
Title: Duplication in Chitotriosidase (CHIT1) Gene and the Risk for Aspergillus Lung Disease in CF Patients.

Introduction: Chitinases are the enzymes that digest the chitin polymer. Plants use CHIT1 as an important innate defense mechanism against fungi. CHIT1 is the major chitinase in the human airways.Variation in the coding region, with 24-bp duplication allele results in a reduced CHIT1 activity. Recently, CHIT1 duplication was found in 6/6 patients with severe asthma and fungal sensitization Aspergillus often persists in the respiratory tract of patients with Cystic Fibrosis (CF) and may cause allergic broncho pulmonary aspergillosis (ABPA).

Aim: to evaluate the link between CHIT1 duplication in CF patients and the predisposition to ABPA or persistent Aspergillus infection.

Patients: 40 CF patients divided to three groups .Group 1: patients who have neither ABPA nor Aspergillus infection in the past (the control group).Group 2: patients with persistent Aspergillus infection, without ABPA. Group 3: patients with current or past ABPA.

Design: Observational, single visit. Methods: All patients will be assessed for pulmonary function tests (PFT), sputum cultures, and blood tests for: CHIT1 duplication, IgE and Eosinophils levels.

Patient's characteristics including demographics, CF mutations, pancreatic status and sweat test will be derived from the charts.

Patients with ABPA as well as Aspergillus infection had also radioallergosorbent test (RAST) for molds, as well as skin prick test for Aspergillus and blood Galactomannan.

The primary outcome measure is the difference in CHIT1 genotyping between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cystic Fibrosis.

Exclusion Criteria:

* Inability to produce sputum, or previous history of lung transplantation.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 40 Cystic Fibrosis patients: Group 1: 22 CF patients who had neither ABPA nor Aspergillus infection in the past.
  Group 2: 12 CF patients with persistent Aspergillus infection, without ABPA. Group 3: 6 CF patients with current or past ABPA
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
CHIT1 genotyping | Baseline
  In peripheral blood.

SECONDARY OUTCOMES:
IgE | Baseline
  peripheral blood count
Eosinophils | Baseline
  peripheral blood count
skin test for aspergillus | Baseline
  skin prick test
galactomannan | Baseline
  peripheral blood count
pulmonary function test | Baseline
  spirometry
RAST test | Baseline
  Radioallergosorbent test (RAST) for molds

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

REFERENCES:
- [Derived] Livnat G, Bar-Yoseph R, Mory A, Dagan E, Elias N, Gershoni R, Bentur L. Duplication in CHIT1 gene and the risk for Aspergillus lung disease in CF patients. Pediatr Pulmonol. 2014 Jan;49(1):21-7. doi: 10.1002/ppul.22749. Epub 2013 Jan 28. PMID 23359515